CLINICAL TRIAL: NCT00000621
Title: Feasibility of Retinoic Acid Treatment in Emphysema (FORTE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Treatment
Other Study IDs: 124
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Emphysema; Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Tretinoin; Isotretinoin

INTERVENTIONS:
Drug: all trans retinoic acid
Drug: 13 cis retinoic acid
Drug: placebo

SUMMARY:
To conduct feasibility studies on the use of retinoids in the treatment of emphysema. Specific objectives are to identify optimal patient populations, retinoids, doses, dosing schedules, routes of administration, and outcome measures preparatory to conducting a larger, controlled, clinical trial on the efficacy of retinoid therapy in the management of emphysema.

DETAILED DESCRIPTION:
BACKGROUND:

Chronic obstructive pulmonary disease (COPD), which includes chronic bronchitis and emphysema, affects more than 16 million Americans, is the fourth leading cause of death in the USA, and costs the nation billions in direct and indirect health care costs. Though only about two million of the 16 million people with COPD have emphysema, emphysema is more disabling, accounting for approximately half of the 114 million days of restricted activity and half of the 53 million days of disability attributed to COPD per year. Emphysema is characterized by destruction of the air space walls, leading anatomically to abnormal, persistent enlargement of the airspaces distal to the terminal bronchioles, and without obvious fibrosis. The clinical result is continuous dyspnea due to hyperinflation of the lung, over distention of the chest wall, disadvantaged respiratory muscles, and hypoxia, even at rest.

Treatment options in emphysema are limited and primarily aimed at symptomatic relief of the dyspnea by maximizing the depleted reserves of the patient. In the late stages, care is supportive, in the form of oxygen therapy, bronchodilator, nutritional supplementation and exercise rehabilitation. Exercise rehabilitation has been shown to improve the quality of life, but only oxygen therapy has been shown to affect survival. For patients less than 60 years old, lung transplantation may be possible, but scarcity of donor lungs and expense greatly limits this option and the efficacy has not been studied. Lung volume reduction surgery is currently under investigation for its effect on symptoms and survival. For the few patients with hereditary alpha-1-antitrypsin deficiency, the recent report of the NHLBI supported Alpha-1-Antitrypsin Deficiency Registry Study Group cautions that although those with moderate airflow obstruction may benefit from augmentation therapy, more studies were needed to draw firm conclusions and to answer questions about dose and dosing schedules.

Recent laboratory data have shown that all-trans-retinoic acid, a derivative of vitamin A, can regenerate alveoli in adult rats with elastase induced emphysema (Massaro, GD and Massaro D. Retinoic Acid Treatment Abrogates Elastase-induced Pulmonary Emphysema in Rats. Nature Med 3:675-677, 1997). Based upon the findings that prior to septation, rats have fibroblasts rich in vitamin A storage granules, high concentrations of cellular retinol binding protein, and lung nuclear retinoic acid binding receptors, all of which diminish after septation and the fact that retinoic acid increases the number of alveoli in rats, the investigators reasoned that retinoic acid plays a key role in septation. Tracheal instillation of elastase into adult rats resulted in an increase in lung volume, a decrease in surface area, and large alveoli as in human emphysema. Intra peritoneal injection of all-trans retinoic acid in the elastase-treated rats for 12 days prior to sacrifice reduced the lung volume and increased the surface area to normal.

In addition to the elastase-treated rats, all trans-retinoic acid has been found to induce formation of alveoli in normal rats, in neonatal rats treated with dexamethasone, which prevents septation, in adult tight skin mice, and in fetal mouse lung in culture.

These findings led to interest in the medical community whether adult emphysema patients might get symptomatic relief from treatment with all-trans-retinoic acid. In September 1998, the NHLBI convened a workshop, entitled "Clinical Trial Feasibility: All-trans-Retinoic Acid for the Treatment of Emphysema", to discuss the feasibility of a clinical trial to test the efficacy of retinoic acid in the treatment of emphysema. The workshop participants agreed that the laboratory findings were exciting, but that a proof of principle study was needed to demonstrate whether the laboratory findings could be applied to humans with emphysema. Since there was adequate information about the dose range and toxicity of retinoids in humans, adequate methods for assessing the extent of emphysema, and adequate methods to assess the biological activity and distribution of retinoids in the human lung, the workshop participants thought studies in emphysema patients were possible and appropriate. Several possible populations and retinoids, especially the retinoic acids, were discussed as appropriate for a clinical trial. However, the participants did not think that there was sufficient information available to recommend a single trial design and recommended the conduct of multiple small trials, allowing flexibility in the choice of population, retinoid, doses, and outcomes.

DESIGN NARRATIVE:

The core study is a multi-center, randomized, double-masked, placebo-controlled clinical trial enrolling a total of 300 non-smoking persons with emphysema at 5 participating clinical centers. Study participants were randomly assigned in a 1:1:1 ratio to one of three retinoid treatment arms. Within each study arm, participants were randomized to active treatment or to a matched placebo in a 3:1 ratio. After six months of follow-up, the three month crossover period began. Participants initially assigned to active treatment began taking the matched placebo, and participants originally assigned placebo began taking the active treatment. Retinoid treatment arms were all-trans retinoic acid (ATRA trademark, Roche Laboratories, Inc.) at two different doses and 13-cis retinoic acid (cRA, Roche Laboratories, Inc.), each with matched placebo. Several single-center substudies were also performed.

ELIGIBILITY:
1. Men and women > 45 years.
2. Women of child-bearing potential must agree to use two forms of contraception or abstinence, and undergo monthly pregnancy testing.
3. No inhaled nicotine for >= 6 months and cotinine < 20 ng/mL.
4. Best FEV1 >= 25% of predicted and <= 80% of predicted on initial screening, using Hankinson's predicted values.
5. DLCO <= 80% predicted on initial screening, using Crapo's predicted values (corrected for hemoglobin).
6. Spiral CT scan evidence of emphysema: visual impression of at least 10% emphysema on a fixed section of the total lung, and at least 10% of the lung with < -910 HU.
7. PCO2 < 45 mm Hg, and willingness to undergo bronchoscopy if FEV1 >= 30% of predicted.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)